CLINICAL TRIAL: NCT05916326
Title: A Phase III Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Protective Efficacy, Safety and Immunogenicity of Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula Polymorpha) in Healthy People Aged 6 Months to 13 Years
Brief Title: Phase III Clinical Trial to Evaluate the Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula Polymorpha)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CXSL1700011-III
Record Dates: First submitted 2023-06-06; First posted 2023-06-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Norovirus Infections; Norwalk Gastroenteritis
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental vaccine group (Experimental)
  Interventions: Biological: Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha)
- placebo group (Placebo Comparator)
  Interventions: Biological: placebo
- Experimental vaccine group（Immunogenic subgroup ） (Experimental)
  Interventions: Biological: Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha)
- placebo group（Immunogenic subgroup） (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) — Intramuscular injection of Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) in the deltoid muscle of the upper arm
  Arms: Experimental vaccine group; Experimental vaccine group（Immunogenic subgroup ）
Biological: placebo — Intramuscular injection of placebo in the deltoid muscle of the upper arm
  Arms: placebo group; placebo group（Immunogenic subgroup）

SUMMARY:
The purpose of this study is to evaluate the Efficacy, Safety and Immunogenicity of the Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) in Healthy People Aged 6 Months to 13 Years After Vaccination

ELIGIBILITY:
Inclusion Criteria:

* Aged from 6 months to 13 years old, and can provide legal identity certificate;
* Volunteers and/or their guardians have the ability to understand the study requirements and process, agree to participate in the clinical trial and sign the informed consent, and can participate in all planned follow-up visits ( by an authorized entrusted person on the premise of written authorization by the guardian the informed consent can be signed);
* Those <12 months old: born in full-term pregnancy (gestational week 37-42 weeks) and birth weight ≥ 2.5kg.

Exclusion Criteria:

First dose exclusion criteria：

* Axillary body temperature > 37.0°C ;
* Have a history of chronic gastrointestinal diseases;
* Had gastroenteritis requiring treatment or current diarrhea, vomiting or other digestive system diseases within 7 days;
* Have a history of allergy to any excipients of the experimental vaccine (L-histidine, sodium chloride, aluminum hydroxide and water for injection, etc.);
* Have a history of severe allergy to any vaccine or drug, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, Arthus reaction;
* Have been diagnosed with congenital or acquired immunodeficiency, or received immunosuppressant treatment, such as the application of systemic glucocorticoid therapy for more than 2 consecutive weeks 2 months before vaccination, such as prednisone or similar drugs > 5mg/day (note: use of topical and inhaled/nebulized steroids can participate);
* Infectious diseases, such as: tuberculosis, viral hepatitis or parents infected with human immunodeficiency virus HIV;
* Thrombocytopenia, any coagulation disorders, or intramuscular injection contraindications receiving anticoagulant therapy etc.;
* The volunteer himself or his biological parents have a history of convulsions (except for febrile convulsions in children), epilepsy and mental illness;
* Serious diseases or congenital malformations that may interfere with the conduct or completion of the research (including but not limited to: asthma and other respiratory diseases or during the attack of chronic bronchitis, Down syndrome, thalassemia, heart disease, encephalopathy, kidney disease, self immune diseases, genetic allergies, Guillain-Barre Syndrome, severe skin diseases, severe malnutrition, severe developmental disorders, etc.);
* Asplenia, functional asplenia, and asplenia or splenectomy caused by any reason;
* Have received blood or blood-related products or immune globulin within 3 months (hepatitis B immune globulin and rabies patient immune globulin are acceptable);
* vaccinated inactivated/recombinant vaccines (non-live vaccines) within 7 days, and inoculate live attenuated vaccines or COVID-19 vaccines within 14 days;
* Acute illness or acute exacerbation of chronic disease within 3 days;
* Have taken antipyretic, analgesic or antiallergic drugs within 3 days;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* Participating in or planning to participate in another interventional research during the study process;
* The investigators believe that the volunteers have other conditions that may interfere with the evaluation of the research purpose;
* <12 months old: the baby is born with abnormal labor process (dystocia, instrumental midwifery) or has a history of suffocation, nervous system damage, current pathological jaundice, perianal abscess, severe eczema;
* If there have been serious adverse reactions after vaccination in the past, the investigator will determine whether the volunteer is enrolled or not according to the actual situation.

If items 1, 3, 13, 14, and 15 of the exclusion criteria are met, the volunteer's enrollment will be postponed.

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8000 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of moderate/severe acute gastroenteritis caused by laboratory-confirmed (RT-PCR) infection with GI.1 or GII.4 norovirus after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14 days after the full course of vaccination to end of study（about two years）
  Efficacy：The sum of the incidence rate of the placebo group and the incidence rate of the experimental group, divided by the incidence rate of the placebo group

SECONDARY OUTCOMES:
To evaluate the efficacy of against moderate/severe acute gastroenteritis caused by laboratory-confirmed (RT-PCR) infection with any strain of norovirus | 14 days after the full course of vaccination to end of study（about two years）
  after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha)
  Efficacy：The sum of the incidence rate of the placebo group and the incidence rate of the experimental group, divided by the incidence rate of the placebo group
To evaluate efficacy of any gastroenteritis caused by laboratory-confirmed (RT-PCR) infection with GI.1 or GII.4 norovirus after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14 days after the full course of vaccination to end of study（about two years）
  Efficacy：The sum of the incidence rate of the placebo group and the incidence rate of the experimental group, divided by the incidence rate of the placebo group
To evaluate the efficacy of any gastroenteritis caused by laboratory-confirmed (RT-PCR) infection with any strain of norovirus after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14 days after the full course of vaccination to end of study（about two years）
  Efficacy：The sum of the incidence rate of the placebo group and the incidence rate of the experimental group, divided by the incidence rate of the placebo group
IgG of NoV GI.1 and GII.4 after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14th day after the full course of vaccination
  only Immunogenic subgroup
HBGA-blocking antibody geometric mean titer (GMT) of NoV GI.1 and GII.4 after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14th day after the full course of vaccination
  only Immunogenic subgroup
Positive conversion rates of GMT for NoV GI.1 and GII.4 after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14th day after the full course of vaccination
  only Immunogenic subgroup
Compared to before vaccination，the growth multiple of GMT for NoV GI.1 and GII.4 antibodies after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 14th day after the full course of vaccination
  only Immunogenic subgroup
HBGA-blocking antibodies Geometric mean titer (GMT) of NoV GI.1 and GII.4 after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 180th,360th,540th,720th day after the full course of vaccination
  only Immunogenic subgroup
IgG of NoV GI.1 and GII.4 after full vaccination with Human Norovirus Bivalent (GⅠ.1/GⅡ.4)Vaccine，Recombinant (Hansenula polymorpha) | 180th,360th,540th,720th day after the full course of vaccination
  only Immunogenic subgroup
the incidence and severity of adverse reactions/events within 30 minutes after each dose of vaccination | The period after each dose to 30 minutes after the dose
the incidence and severity of adverse reactions/events within 0-7 days after each dose of vaccination | The period after each dose to 7 days after the dose
the incidence and severity of non-solicited adverse reactions/events within 28 days after each dose of vaccination | The period after each dose to 28 days after the dose
the incidence of SAE from the first dose of vaccination to end of study | the first dose of vaccination to end of study（about two years）

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Laishui County Center for Disease Control and Prevention, Baoding, Hebei
  - Jingxing County Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Zhao County Center for Disease Control and Prevention, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No